CLINICAL TRIAL: NCT05599841
Title: Evaluation of the Systemic Effect of Intraoperative Diluted Povidone Iodine Irrigation Using Urine Iodine and Thyroid Function Tests in Patients Undergoing Knee-Hip Arthroplasty
Brief Title: Povidone Iodine Irrıgation at Hip-Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Hakan KOCAOGLU, M.D. Assoc. Prof., Ankara University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: Orthop2180
Record Dates: First submitted 2022-10-26; First posted 2022-10-31 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Osteoarthritis; Hyperthyroidism; Iodine Toxicity
MeSH Terms: conditions — Osteoarthritis; Hyperthyroidism | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Povidone Iodine Solution (Active Comparator): The group whom PI solution will be used at surgery
  Interventions: Procedure: PI solution
- Saline Solution (Placebo Comparator): The group whom only saline solution will be used at surgery
  Interventions: Procedure: Saline Solution

INTERVENTIONS:
Procedure: PI solution — 3,000 cc of <2% concentrated povidone iodine solution will be used as irrigation solution at primary hip/knee arthroplasty. The PI solution was left in the joint for 3 minutes.
  Arms: Povidone Iodine Solution
Procedure: Saline Solution — 3,000 cc of 0.9% saline solution will be used as irrigation solution at primary hip/knee arthroplasty. The saline solution was left in the joint for 3
  Arms: Saline Solution

SUMMARY:
Povidone iodine (PI) solution is an antimicrobial solution that can be used at hip and knee arthroplasty cases. It contains iodine that may be absorbed by the body. This study aims to investigate any absorption caused by PI solution.

ELIGIBILITY:
Inclusion Criteria:

* All patients with hip/knee osteoarthritis who undergo primary arthroplasty

Exclusion Criteria:

* Patients with abnormal thyroid function tests in the preoperative period, a history of the previous thyroid-related disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-09-16 (Estimated)

PRIMARY OUTCOMES:
Urine iodine level | postoperative first day
  Urine iodine concentration

SECONDARY OUTCOMES:
Thyroid hormone | postoperative 14 days
  Blood thyroid hormone levels including: TSH, T3 and T4

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Kocaoglu, MD, Principal Investigator — Ankara University
Locations (1):
- Ankara University Faculty of Medicine, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ertan MB, Basarir K, Kocaoglu H, Aydugan MY, Gungor E. Systemic iodine levels increase with povidone-iodine irrigation, but does this affect thyroid functions? A case-control study. J Orthop Surg Res. 2024 Oct 8;19(1):636. doi: 10.1186/s13018-024-04877-8. PMID 39380015